CLINICAL TRIAL: NCT00379080
Title: A Feasibility Assessment and a Phase I/II Trial of MLN518 for Treatment of Patients With Recurrent Glioblastoma
Brief Title: Tandutinib in Treating Patients With Recurrent or Progressive Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00681; NCI-2009-00681 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000495253; NABTT 0504 (Other: Adult Brain Tumor Consortium); NABTT-0504 (Other: CTEP); U01CA137443 (NIH)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Adult Brain Tumor; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — tandutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I - Feasibility (Experimental): Patients receive oral tandutinib twice daily for 7 days. Patients then undergo biopsy or surgery to remove the tumor. Within 2 weeks after biopsy or surgery, patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  conventional surgery
  oral tandutinib
  Pharmacological study
  Tissue samples
  Interventions: Procedure: conventional surgery; Drug: tandutinib; Other: pharmacological study; Other: Tissue samples
- Arm 2 - Dose Escalation (Phase 1) (Experimental): Phase I: Patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of tandutinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.
  the starting dose for tandtinib is 500mg BID
  oral tandutinib
  Pharmacological study
  Tissue samples
  Interventions: Drug: tandutinib; Other: pharmacological study; Other: Tissue samples
- Arm 3 - Phase 2 (Experimental): Patients receive tandutinib as in phase I at the MTD determined in phase I.
  600mg was the determined MTD in Dose Escalation
  oral tandutinib
  Pharmacological study
  Tissue samples
  Interventions: Drug: tandutinib; Other: pharmacological study; Other: Tissue samples

INTERVENTIONS:
Procedure: conventional surgery — Undergo surgery
  Other Names: MLN518
  Arms: Arm I - Feasibility
Drug: tandutinib — Given orally
  Other Names: CT53518
Other: pharmacological study — Correlative studies
Other: Tissue samples — Correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of tandutinib and to see how well it works in treating patients with recurrent or progressive glioblastoma.Tandutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the ability of tandutinib to achieve a target tumor/plasma ratio ≥ 0.33 in patients with recurrent glioblastoma undergoing resection. (Feasibility study) II. Detect potential biological effects of tandutinib by measuring platelet-derived growth factor receptor phosphorylation status and downstream activation of Akt and Erk. (Feasibility study) III. Determine the maximum tolerated dose of tandutinib in patients with recurrent or progressive glioblastoma. (Phase I) IV. Estimate the frequency of toxicities associated with tandutinib in patients with recurrent or progressive glioblastoma. (Phase I) V. Describe the pharmacokinetics of this route of administration in patients with recurrent or progressive glioblastoma. (Phase I) VI. Assess tumor response rate in patients with recurrent or progressive glioblastoma. (Phase II)

SECONDARY OBJECTIVES:

I. Estimate overall survival of patients with recurrent or progressive glioblastoma. (Phase II) II. Estimate the 6-month progression-free survival rate in these patients. (Phase II) III. Assess the toxicities associated with tandutinib in these patients. (Phase II) IV. Assess the pharmacokinetic profile of this route of administration in these patients. (Phase II) V. Explore protein-expression patterns that distinguish patients who respond to therapy from those who do not. (Phase II)

OUTLINE: This is a multicenter, prospective, nonrandomized, feasibility study and phase I study (in parallel) followed by an open label phase II study.

FEASIBILITY STUDY: Patients receive oral tandutinib twice daily for 7 days. Patients then undergo biopsy or surgery to remove the tumor. Within 2 weeks after biopsy or surgery, patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE I: Patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of tandutinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

[Note: *On day 1 of course 1, patients receive only 1 dose of tandutinib.]

PHASE II: Patients receive tandutinib as in phase I at the MTD determined in phase I.

Patients undergo blood sample collection for pharmacokinetic studies. Patients in the feasibility portion of the study also undergo blood and tissue sample collection for correlative studies by mass spectrometry for tandutinib concentration. Samples are also examined for circulating endothelial cells and plasma proteins (vascular endothelial growth factor [VEGF]-A, -B, -C, and -D, soluble VEGF receptors [sVEGFR's], placental growth factor [P1GF], platelet-derived growth factor [PDGF]-AA, PDGF-AB, PDGF-BB, angiopoietin-1 and -2, tumstatin, thrombospondin-1, and IL-8) as potential markers of the antiangiogenic effect of tandutinib.

After completion of study treatment, patients are followed every 2 months.

ELIGIBILITY:
Criteria:

* Histologically confirmed glioblastoma:

  * Progressive or recurrent disease after prior radiotherapy (with or without chemotherapy)
  * Patients with a previous low-grade glioma that progressed after prior radiotherapy (with or without chemotherapy) and are found to have glioblastoma by biopsy are eligible
* Measurable disease, defined as contrast-enhancing progressive or recurrent glioblastoma by MRI or CT imaging within the past 2 weeks
* Must be maintained on a stable corticosteroid regimen from the time of baseline scan to the start of study treatment
* Feasibility study only:

  * Planning to undergo surgical resection or biopsy
  * Stereotactic biopsy for confirmation of tumor progression or differentiation of tumor progression from treatment-induced effects allowed
  * Corticosteroids must be tapered to the lowest required steroid dose and patient must be maintained on a stable dose after surgery or biopsy
* Karnofsky performance status 60-100%
* Absolute neutrophil count >= 1,500/mm^3
* Hemoglobin >= 10 mg/dL
* Bilirubin =< 1.5 mg/dL
* AST and ALT =< 4 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier method contraception during and for 3 months after completion of study treatment
* Mini Mental State Exam score >= 15
* Mean QTc =< 500 msec (with Bazett's correction) by screening electrocardiogram
* LVEF >= 40%
* No history of familial long QT syndrome
* No myocardial infarction within the past 6 months
* No severe uncontrolled ventricular arrhythmias
* No uncontrolled angina
* No electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* No ongoing vomiting or nausea >= grade 2
* No gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous alimentation
* No active peptic ulcer disease
* No other condition that would impair ability to swallow pills or absorb oral medications
* No muscular dystrophy
* No myasthenia gravis
* No other known or suspected primary muscular or neuromuscular disease
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to tandutinib (e.g., erlotinib hydrochloride, gefetinib, or doxazosin mesylate)
* Patients who developed an acneiform/maculopustular rash while receiving either gefitinib or erlotinib hydrochloride are eligible unless the rash is considered an allergic reaction (angioedema/urticaria) or Stevens-Johnson syndrome
* No ongoing or active infections
* No psychiatric illness or social situations that would preclude study compliance
* No other serious infection or medical illness
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No other uncontrolled illness
* No other malignancy within the past 5 years except for basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* Recovered from prior therapy
* At least 3 months since prior radiotherapy
* No prior surgical procedures affecting absorption
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No concurrent agent that would cause QTc prolongation
* No concurrent prophylactic growth factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])
* At least 10 days since prior and no concurrent anticonvulsant drugs that induce hepatic metabolic enzymes (e.g., primidone, oxcarbazepine, phenytoin, carbamazepine, or phenobarbital)
* No prior treatment with small molecule inhibitors of platelet-derived growth factor receptor (e.g., sunitinib malate, sorafenib, or imatinib mesylate)
* Platelet count >= 100,000/mm^3
* No New York Heart Association class III or IV heart failure
* Creatinine =< 1.5 mg/dL OR creatinine clearance >= 60mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-01; Primary Completion 2012-09 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Batchelor, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from 4/2007 through 6/2010. Patients accrued in the outpatient clinical setting. The first part of study was for patients who required surgery. Hence these patients were treated in-patient.
Groups:
- Arm 1- Phase 0: Patients receive oral tandutinib twice daily for 7 days. Patients then undergo biopsy or surgery to remove the tumor. Within 2 weeks after biopsy or surgery, patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  conventional surgery
  oral tandutinib
  Pharmacological study
  Tissue samples
- Arm 2 - Phase 1: Phase I: Patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  tandutinib: Given orally
  pharmacological study: Correlative studies
- Arm 3 - Phase 2: Patients receive tandutinib as in phase I at the MTD determined in phase I.
  600mg was the determined MTD in Dose Escalation
  oral tandutinib
  Pharmacological study
  Tissue samples
  tandutinib: Given orally
  pharmacological study: Correlative studies
  Tissue samples: Correlative studies
Period: Overall Study
Arm/Group | Arm 1- Phase 0 | Arm 2 - Phase 1 | Arm 3 - Phase 2
Started | 6 | 19 | 31
Completed | 6 | 15 | 31
Not Completed | 0 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Population: all pts had to have confirmed histological GBM, prior treatment wih RT and a MMSE of greater or equal to 15.
Groups:
- Arm 1 - Phase 0: Patients receive oral tandutinib twice daily for 7 days. Patients then undergo biopsy or surgery to remove the tumor. Within 2 weeks after biopsy or surgery, patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  conventional surgery
  oral tandutinib
  Pharmacological study
  Tissue samples
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Phase 0 | Arm 2 - Phase 1 | Arm 3 - Phase 2 | Total
Number analyzed (Participants) | 6 | 19 | 31 | 56
Age, Continuous [Median (Full Range); unit: years] | 61 [48 to 72] | 56 [42 to 77] | 54 [24 to 69] | 56 [24 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 7 | 13
  Male | 4 | 15 | 24 | 43
Karnofsky Performance Status [Median (Full Range); unit: Percentage] — Higher score better 100 normal no complaints/disease 90 capable normal activity few symptoms/disease 80 normal activity, some difficulty some symptoms/signs 70 caring for self not capable normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  Percentage | 80 [60 to 100] | 90 [60 to 100] | 90 [60 to 100] | 90 [60 to 100]
Mini Mental Score [Median (Full Range); unit: units on a scale] — The mini-mental state examination (MMSE) is a 30-point questionnaire test used to screen for cognitive impairment. Commonly used to screen for dementia. It is also used to estimate the severity of cognitive impairment and to follow the course of cognitive changes in an individual over time. The MMSE test includes simple questions and problems in a number of areas: the time and place of the test, repeating lists of words, arithmetic such as the serial sevens, language use and comprehension, and basic motor skills. The Higher your score, the higher your function. Scale Ranges from 1-30
  units on a scale | 29 [20 to 30] | 30 [22 to 30] | 29 [15 to 30] | 29 [15 to 30]
Steroids [Number; unit: participants]
  Yes | 5 | 10 | 8 | 23
  No | 1 | 9 | 23 | 33

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Tandutinib Defined by Dose Limiting Toxicities (Phase 1)
Time Frame: cycle 1 - 28 days
Population: 19 patients enrolled in dose escalation but 4 were removed for reasons other than drug related toxicity
Measure: Number; unit: mg BID
Groups:
- Reporting Group - Phase 1: Phase I: Patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. All dose Levels
  tandutinib: Given orally
  pharmacological study: Correlative studies
Arm/Group | Reporting Group - Phase 1
Number analyzed (Participants) | 15
mg BID | 600

2. Primary Outcome: To Determine the Tumor/Plasma Ratio of in Subjects With Recurrent GBM Undergoing Resections (Phase 0)
Description: participants are administered tandutinib (500mg BID) for 7 days prior to surgery and then undergo resection for recurrent glioblastoma. Tissue samples will be collected for correlative studies - determine tumor/plasma ratio.
Time Frame: 7 days prior to surgery including surgery
Population: a tandutinib tumor:plasma ratio of >/=0.33 was the objective in a minimum of 3/6 subjects in order to proceed with Phase 1/2 study. 6 samples received, but 2 samples were found to be thawed at receipt and not used in analysis
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Arm I - Feasibility: Participants receive oral tandutinib 500 mg twice daily for 7 days prior to surgery. Patients then undergo biopsy or surgery to remove the tumor. Tissue collected for tumor/plasma ratio.
  Post surgery, within 2 weeks after biopsy or surgery, patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. (not necessary for feasibility)
  conventional surgery
  oral tandutinib
  Pharmacological study
  Tissue samples
  conventional surgery: Undergo surgery
  tandutinib: Given orally
  pharmacological study: Correlative studies
  Tissue samples: Correlative studies
Arm/Group | Arm I - Feasibility
Number analyzed (Participants) | 4
ratio | 13.1 (8.9)

3. Primary Outcome: Number of Dose Limiting Toxicities Per Dose Level
Description: cohorts of 3-6 pts will recieve oral tandutinib starting at 500mg BID with a dose escalation in each cohort. Each treatment cycle is 28 days. Evaluation period for MTD is 1st cycle - 28 days.
  dose limiting toxicity defined as: grades 3-4 severity (except vomiting and diarrhea without sufficient prophylaxis delay of treatment > 14 days. ANC less/equal 500m/mm3; Plts less/equal 25,000/mm3; febrile neutropenia or delay of treatment > 14 days
Time Frame: 28 days
Population: all GBM, All prior treatment with RT. assessment was for 28 days, cycle 1. 3 dose levels 500, 600 and 700mg
Measure: Number; unit: participants
Groups:
- Level 1 - 500mg BID: Phase I: Patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of tandutinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.
  dose for tandtinib is 500mg BID
  oral tandutinib
  Pharmacological study
  Tissue samples
  tandutinib: Given orally
  pharmacological study: Correlative studies
  Tissue samples: Correlative studies
- Level 2 - 600mg BID: Phase I: Patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of tandutinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.
  dose for tandtinib is 600mg BID
  oral tandutinib
  Pharmacological study
  Tissue samples
  tandutinib: Given orally
  pharmacological study: Correlative studies
  Tissue samples: Correlative studies
- Level 3 - 700mg BID: Phase I: Patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of tandutinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.
  dose for tandtinib is 700mg BID
  oral tandutinib
  Pharmacological study
  Tissue samples
  tandutinib: Given orally
  pharmacological study: Correlative studies
  Tissue samples: Correlative studies
Arm/Group | Level 1 - 500mg BID | Level 2 - 600mg BID | Level 3 - 700mg BID
Number analyzed (Participants) | 6 | 6 | 3
participants | 1 | 1 | 2

4. Primary Outcome: Tumor Response (Complete Response and Partial Response) Rate (Phase II)
Description: pts receive a scan baseline and prior to every odd cycle. All responses are centrally reviewed Complete response Complete disappearance of all tumor on MRI scan, off all glucocorticoids with stable or improving neurological exam minimum of 4 wks Partial response Greater than or equal 50% reduction in tumor size on MRI, on sable or decreasing glucocorticoids with stable or improving neurological exam for a minimum of 4 wks.
  Progressive disease Progressive neurological abnormalities not explained by other causes or greater than 25% increase in size of tumor or if new lesion.
  Stable disease Clinical status and MRI does not qualify for complete response, partial response or progression
Time Frame: Up to 4 years
Population: In the first stage, 31 patients would be enrolled and the trial would be terminated if 3 or fewer patients demonstrated objective responses (partial response or complete response)
Measure: Number; unit: participants with objective response
Arm/Group | Arm 3 - Phase 2
Number analyzed (Participants) | 31
participants with objective response | 1

5. Primary Outcome: Pharmacokinetics (Max Concentration of Plasma) for Tandutinib in Phase 1 and Phase 2
Description: pre-dose, 1,2,4,6,8 and 24 hrs post dose and days 8,15, 21 of cycle 1 and day one of cycle 2
Time Frame: 28 days
Population: 56 enrolled pts, 40 evaluable PK sample sets, parameters not estimated for 16 pts. (Sample collected after next dose taken 3pts;1st dose given before collecting redose sample 1 pt; concentration sample 24h after dosing <LOQ 8 pts or samples not collected proper times 1pt. 2pts feasibility arm did not restart treatment post-surgery
Measure: Median (Standard Deviation); unit: ng/mL
Groups:
- Level 2 - 600mg BID (Phase 1 & Phase 2): Phase I: Patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of tandutinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.
  Phase 2: MTD dose Patients receive tandutinib as in phase I at the MTD (600mg BID) determined in phase I.
  600mg was the determined MTD in Dose Escalation
  dose for tandtinib is 600mg BID
  oral tandutinib
  Pharmacological study
  Tissue samples
  tandutinib: Given orally
  pharmacological study: Correlative studies
  Tissue samples: Correlative studies
Arm/Group | Level 1 - 500mg BID | Level 2 - 600mg BID (Phase 1 & Phase 2) | Level 3 - 700mg BID
Number analyzed (Participants) | 6 | 31 | 3
ng/mL | 379 (193) | 486 (307) | 1285 (239)

6. Primary Outcome: Pharmacokinetics (Apparent Terminal Phase Half-life) for Tandutinib in Phase 1 and Phase 2
Description: pre-dose, 1,2,4,6,8 and 24 hrs post dose and days 8,15, 21 of cycle 1 and day one of cycle 2
Time Frame: 28 days
Population: as for outcome 5
Measure: Median (Standard Deviation); unit: h
Groups:
- Level 2 - 600mg BID: Phase I: Patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of tandutinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.
  Phase 2: MTD dose Patients receive tandutinib as in phase I at the MTD (600mg BID) determined in phase I.
  600mg was the determined MTD in Dose Escalation
  dose for tandtinib is 600mg BID
  oral tandutinib
  Pharmacological study
  Tissue samples
  tandutinib: Given orally
  pharmacological study: Correlative studies
  Tissue samples: Correlative studies
Arm/Group | Level 1 - 500mg BID | Level 2 - 600mg BID | Level 3 - 700mg BID
Number analyzed (Participants) | 6 | 31 | 3
h | 13.1 (1.1) | 10.4 (2.5) | 13.2 (7.2)

7. Primary Outcome: Pharmacokinetics (Area Under the Plasma Concentration Time Profile From Zero to Infinity (AUC)) for Tandutinib in Phase 1 and Phase 2
Description: pre-dose, 1,2,4,6,8 and 24 hrs post dose and days 8,15, 21 of cycle 1 and day one of cycle 2
Time Frame: 28 days
Population: as for outcome 5
Measure: Median (Standard Deviation); unit: ng*h/mL
Arm/Group | Level 1 - 500mg BID | Level 2 - 600mg BID | Level 3 - 700mg BID
Number analyzed (Participants) | 6 | 31 | 3
ng*h/mL | 3961 (1414) | 4659 (1926) | 8193 (1915)

8. Primary Outcome: Pharmacokinetics; Apparent Oral Clearance for Tandutinib in Phase 1 and Phase 2
Description: pre-dose, 1,2,4,6,8 and 24 hrs post dose and days 8,15, 21 of cycle 1 and day one of cycle 2
Time Frame: 28 days
Population: 56 enrolled pts, 40 evaluable PK sample sets, parameters not estimated for 16 pts. (Sample collected after next dose taken 3pts;1st dose given before collecting redose sample 1 pt; concentration sample 24h after dosing <LOQ 8 pts or samples not collected proper times 1pt. 2pts feasibility arm did not restart treatment post surgery
Measure: Median (Standard Deviation); unit: L/h
Arm/Group | Level 1 - 500mg BID | Level 2 - 600mg BID | Level 3 - 700mg BID
Number analyzed (Participants) | 6 | 31 | 3
L/h | 126 (45) | 129 (54) | 85 (20)

9. Primary Outcome: Pharmacokinetics; Apparent Oral Total Body Volume of Distribution for Tandutinib in Phase 1 and Phase 2
Description: pre-dose, 1,2,4,6,8 and 24 hrs post dose and days 8,15, 21 of cycle 1 and day one of cycle 2
Time Frame: 28 days
Population: as for outcome 5
Measure: Median (Standard Deviation); unit: L
Arm/Group | Level 1 - 500mg BID | Level 2 - 600mg BID | Level 3 - 700mg BID
Number analyzed (Participants) | 6 | 31 | 3
L | 2386 (934) | 1987 (1102) | 1764 (1242)

10. Primary Outcome: Pharmacokinetics; Steady-state Trough Concentration for Tandutinib in Phase 1 and Phase 2
Description: pre-dose, 1,2,4,6,8 and 24 hrs post dose and days 8,15, 21 of cycle 1 and day one of cycle 2
Time Frame: 28 days
Population: as for outcome 5
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | Level 1 - 500mg BID | Level 2 - 600mg BID | Level 3 - 700mg BID
Number analyzed (Participants) | 6 | 31 | 3
ng/mL | 518 (182) | 582 (381) | 971 (729)

11. Secondary Outcome: Overall Survival (Phase II)
Description: Median time of survival along with 95% confidence interval will be estimated using Kaplan-Meier method. An overall failure rate will be estimated with 95% CI.
Time Frame: Up to 4 years
Population: Median time of survival along with 95% confidence interval will be estimated using Kaplan-Meier method. An overall failure rate will be estimated with 95% CI. The overall failure rate is expressed as hazard of failure per person-year of follow-up.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 3 - Phase 2
Number analyzed (Participants) | 31
months | 8.8 [5.9 to 15.4]

12. Secondary Outcome: Six-month Progression-free Survival Rate (Phase II)
Description: The probability of 6-momth progression-free survival will be estimated using binomial distribution.
  Progression defined as: Progressive neurological abnormalities not explained by other causes or greater than 25% increase in size of tumor or if new lesion.
Time Frame: At 6 months
Population: The probability of 6-momth progression-free survival will be estimated using binomial distribution.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Arm 3 - Phase 2
Number analyzed (Participants) | 31
percent probability | 16 [6 to 34]

13. Secondary Outcome: Overall Failure Rate (Phase II)
Description: The overall failure rate is expressed as hazard of failure per person-year of follow-up.
Time Frame: up to 4 years
Measure: Number (95% Confidence Interval); unit: failure per person-year
Arm/Group | Arm 3 - Phase 2
Number analyzed (Participants) | 31
failure per person-year | 0.82 [0.57 to 1.19]

14. Secondary Outcome: Proportion of Patients With Serious or Life Threatening Toxicities
Description: Grade 3 or 4 toxicities related to treatment as determined by the CTCAE
Time Frame: 2 year period
Measure: Number; unit: percentage of participants
Arm/Group | Arm 3 - Phase 2
Number analyzed (Participants) | 31
percentage of participants | 48

15. Secondary Outcome: Protein Expression Patterns Post Treatment - Loss or Gain
Description: serial blood samples over multiple time points (prior to treatment, 2 days post treatment, 8 days post treatment, 10 days post treatment and 28 days post treatment.
  statistical analyses presented for the comparisons that yielded a p-value <=0.05
Time Frame: baseline - cycle 2 (28 days)
Population: peripheral blood was obtained from 20 patients enrolled in the phase 2 portion of the study.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Groups:
- Baseline (BL) - Overall Survival (OS); Baseline (BL) - Progression Free Survival (PFS); Association Between OS and Biomarker Day 2 / BL; Association Between PFS Biomarker Day 2 / BL; Association Between OS and Biomarker Day 8 / BL; Association Between PFS Biomarker Day 8 / BL; Association Between OS and Biomarker Day 10 /BL; Association Between PFS Biomarker Day 10 / BL; Association Between OS and Biomarker Day 28 / BL; Association Between PFS Biomarker Day 28 / BL: Patients receive tandutinib at 600mg as was the determined MTD in Dose Escalation
  oral tandutinib
  tandutinib: Given orally
  pharmacological study: Correlative studies
  Peripheral blood
Arm/Group | Baseline (BL) - Overall Survival (OS) | Baseline (BL) - Progression Free Survival (PFS) | Association Between OS and Biomarker Day 2 / BL | Association Between PFS Biomarker Day 2 / BL | Association Between OS and Biomarker Day 8 / BL | Association Between PFS Biomarker Day 8 / BL | Association Between OS and Biomarker Day 10 /BL | Association Between PFS Biomarker Day 10 / BL | Association Between OS and Biomarker Day 28 / BL | Association Between PFS Biomarker Day 28 / BL
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 19 | 19 | 18 | 18 | 14 | 14
hazard ratio
  SDF_1a: number analyzed (Participants) | 20 | 20 | 19 | 19 | 17 | 17 | 11 | 11 | 13 | 13
  SDF_1a | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 0.01 [0 to 1.8] | 0.14 [0 to 20] | 0.83 [0.01 to 62] | 0.08 [0 to 24] | 1.4 [0 to 2531] | 1.68 [0 to 3976] | 0.18 [0 to 8.42] | 0.76 [0.02 to 36]
  bFGF: number analyzed (Participants) | 20 | 20 | 19 | 19 | 17 | 17 | 11 | 11 | 14 | 14
  bFGF | 1.00 [0.99 to 1.01] | 1.01 [1.00 to 1.02] | 0.72 [0.42 to 1.23] | 0.52 [0.27 to 1.04] | 1.03 [0.61 to 1.74] | 0.88 [0.53 to 1.47] | 0.65 [0.36 to 1.17] | 0.60 [0.31 to 1.14] | 0.84 [0.44 to 1.61] | 0.70 [0.37 to 1.30]
  PIGF: number analyzed (Participants) | 20 | 20 | 19 | 19 | 17 | 17 | 11 | 11 | 14 | 14
  PIGF | 1.00 [0.99 to 1.01] | 1.01 [1.00 to 1.02] | 8.56 [0.16 to 449] | 1.53 [0.01 to 197] | 3.76 [0.55 to 26] | 11.8 [1.08 to 129] | 0.91 [0.03 to 27] | 0.69 [0.02 to 22] | 1.18 [0.03 to 55] | 6.24 [0.07 to 542]
  sFLT_1: number analyzed (Participants) | 20 | 20 | 19 | 19 | 17 | 17 | 11 | 11 | 14 | 14
  sFLT_1 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 1.08 [0.08 to 1.45] | 1.22 [0.89 to 1.66] | 1.03 [0.86 to 1.23] | 1.12 [0.92 to 1.36] | 1.06 [0.08 to 1.41] | 1.13 [0.82 to 1.55] | 61.5 [1 to 3774] | 524 [4 to 71128]
  VEGF: number analyzed (Participants) | 20 | 20 | 19 | 19 | 17 | 17 | 11 | 11 | 14 | 14
  VEGF | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 0.55 [0.07 to 4.1] | 0.71 [0.12 to 4.14] | 0.43 [0.08 to 2.37] | 0.31 [0.05 to 1.85] | 0.88 [0.34 to 2.26] | 0.74 [0.33 to 1.62] | 1.11 [0.17 to 7.35] | 1.67 [0.2 to 13.7]
  CAIX: number analyzed (Participants) | 19 | 19 | 18 | 18 | 16 | 16 | 11 | 11 | 12 | 12
  CAIX | 1.00 [1.00 to 1.01] | 1.00 [1.00 to 1.00] | 1.16 [0.23 to 5.85] | 0.38 [0.05 to 3.19] | 1.53 [0.99 to 2.36] | 1.74 [1.11 to 2.72] | 1.24 [0.76 to 2.01] | 0.80 [0.44 to 1.45] | 1.41 [0.83 to 2.41] | 0.89 [0.53 to 1.48]
  VEGFR2: number analyzed (Participants) | 20 | 20 | 19 | 19 | 17 | 17 | 12 | 12 | 13 | 13
  VEGFR2 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 0.32 [0.01 to 13.9] | 0.74 [0.02 to 31] | 2.02 [0.07 to 62] | 0.65 [0.02 to 17.3] | 0.10 [0 to 70] | 0.27 [0 to 30] | 0.001 [0 to 1.18] | 0.001 [0 to 0.88]
  ANG_2: number analyzed (Participants) | 20 | 20 | 19 | 19 | 17 | 17 | 12 | 12 | 13 | 13
  ANG_2 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 0.54 [0.04 to 7.42] | 2.15 [0.14 to 33] | 0.89 [0.30 to 2.68] | 1.12 [0.31 to 4.09] | 0.55 [0.13 to 2.36] | 1.05 [0.26 to 4.19] | 0.43 [0.06 to 2.91] | 0.52 [0.05 to 4.93]
Statistical Analysis 1: Comparison: Baseline (BL) - Overall Survival (OS); VEGFR2; Test type: Other; p = 0.04, Regression, Cox
Statistical Analysis 2: Comparison: Association Between PFS Biomarker Day 8 / BL; PIGF; Test type: Other; p = 0.04, Regression, Cox
Statistical Analysis 3: Comparison: Association Between PFS Biomarker Day 8 / BL; CAIX; Test type: Other; p = 0.02, Regression, Cox
Statistical Analysis 4: Comparison: Association Between OS and Biomarker Day 28 / BL; sFLT_1; Test type: Other; p = 0.05, Regression, Cox
Statistical Analysis 5: Comparison: Association Between PFS Biomarker Day 28 / BL; sFLT_1; Test type: Other; p = 0.01, Regression, Cox
Statistical Analysis 6: Comparison: Association Between PFS Biomarker Day 28 / BL; VEGFR2; Test type: Other; p = 0.05, Regression, Cox

ADVERSE EVENTS:
Time Frame: Time of first dose until patient went off treatment. <4 years
Groups:
- Arm I - Feasibility: Patients receive oral tandutinib twice daily for 7 days. Patients then undergo biopsy or surgery to remove the tumor. Within 2 weeks after biopsy or surgery, patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  conventional surgery
  oral tandutinib
  Pharmacological study
  Tissue samples
  conventional surgery: Undergo surgery
  tandutinib: Given orally
  pharmacological study: Correlative studies
  Tissue samples: Correlative studies
- Arm 2 - Dose Escalation (Phase 1): Phase I: Patients receive oral tandutinib twice daily* on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of tandutinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.
  the starting dose for tandtinib is 500mg BID
  oral tandutinib
  Pharmacological study
  Tissue samples
  tandutinib: Given orally
  pharmacological study: Correlative studies
  Tissue samples: Correlative studies
Arm/Group | Arm I - Feasibility | Arm 2 - Dose Escalation (Phase 1) | Arm 3 - Phase 2
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/15 | 15/31
Other Adverse Events (participants affected / at risk) | 3/6 | 15/15 | 28/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Feasibility (N=6) | Arm 2 - Dose Escalation (Phase 1) (N=15) | Arm 3 - Phase 2 (N=31)
confusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
fatigue (General disorders) | 2 (2) | 1 (1) | 3 (3)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 5 (6)
somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
alanine aminotransferase increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 6 (8)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Feasibility (N=6) | Arm 2 - Dose Escalation (Phase 1) (N=15) | Arm 3 - Phase 2 (N=31)
fatigue (General disorders) | 2 (3) | 6 (8) | 14 (18)
Platelet count decrease (Investigations) | 2 (5) | 2 (2) | 6 (20)
anemia (Blood and lymphatic system disorders) | 0 (0) | 4 (19) | 11 (74)
electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 3 (4) | 9 (19)
diarrhea (Gastrointestinal disorders) | 0 (0) | 15 (19) | 19 (37)
nausea (Gastrointestinal disorders) | 0 (0) | 12 (16) | 19 (26)
vomiting (Gastrointestinal disorders) | 0 (0) | 7 (12) | 14 (17)
edema face (General disorders) | 0 (0) | 3 (3) | 6 (7)
edema limb (General disorders) | 0 (0) | 3 (3) | 5 (7)
alanine aminotransferase increased (Investigations) | 0 (0) | 2 (7) | 10 (23)
aspartate aminotransferase increased (Investigations) | 0 (0) | 5 (10) | 8 (23)
white blood cell decreased (Investigations) | 0 (0) | 4 (10) | 11 (45)
creatinine increased (Investigations) | 0 (0) | 1 (3) | 3 (4)
hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 2 (3)
hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6) | 15 (37)
muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
rash maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
blood bilirubin increase (Investigations) | 0 (0) | 2 (2) | 2 (2)
neutrophil count decrease (Investigations) | 0 (0) | 2 (2) | 4 (12)
alkaline phosphatase increase (Investigations) | 0 (0) | 0 (0) | 5 (9)
blurred vision (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 5 (6)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (13)
insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Simon's two-stage design Phase 2, prespecified goal patients alive & progression-free survival 6-months not achieved first stage, 2nd stage not done & trial closed/stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less